CLINICAL TRIAL: NCT01225796
Title: Randomized Trial of Sodium Bicarbonate in Renal Transplant Recipients With Low-normal Serum Bicarbonate Levels
Brief Title: Study of Sodium Bicarbonate in Kidney Transplant Recipients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kalani Raphael, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00044216
Record Dates: First submitted 2010-10-15; First posted 2010-10-21 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Transplantation
Keywords: Bicarbonate; Chronic allograft nephropathy; Urinary TGF-beta; Urinary acid excretion
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium bicarbonate (Experimental): This group will receive oral sodium bicarbonate 650mg three times daily for 6 months.
  Interventions: Drug: Sodium bicarbonate
- Control (No Intervention): This group will not receive any sodium bicarbonate.

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate 650mg by mouth three times daily for 6 months.
  Arms: Sodium bicarbonate

SUMMARY:
The purpose of this study is to compare the effect of sodium bicarbonate versus no sodium bicarbonate treatment on urinary ammonia levels and urinary transforming growth factor-beta1 (TGF-beta1) excretion in renal transplant patients with low-to-normal serum bicarbonate levels (20 - 28 mmol/L).

DETAILED DESCRIPTION:
Renal allograft survival ten years after transplant is only about 50%. In people with non-transplant chronic kidney disease (CKD), sodium bicarbonate treatment seems to delay progressive decline in kidney function in those with low serum bicarbonate levels (metabolic acidosis). This may be because sodium bicarbonate reduces renal ammonia production and hence fibrosis. Observational evidence suggests that people with CKD and low-normal serum bicarbonate levels might also benefit from sodium bicarbonate treatment. TGF-beta1 levels seem to be an important predictor of chronic allograft nephropathy, and alkalinizing agents may have an effect on TFG-beta1 excretion.

Retrospective analysis of participants in the African American Study of Kidney Disease and Hypertension showed the lowest risk of CKD progression was among those having baseline serum bicarbonate levels in the range of 28-30 mmol/L. Recent studies in people with pre-transplant CKD have suggested that increasing low serum bicarbonate levels (< 22 mmol/L) with alkalinizing agents such as sodium bicarbonate and sodium citrate may reduce CKD progression.

Design: this is an open-label randomized study testing the effect of a six-month intervention with sodium bicarbonate 650 mg orally thrice daily versus no sodium bicarbonate treatment on renal ammonia excretion and urinary TGF-beta1.

Visits will occur at baseline, 3 months, and 6 months. At each follow-up visit, the study coordinator or principal investigator will review a medical questionnaire with the participant and collect a sample of blood and urine for analysis of urinary TGF-beta1, metabolic panel, pH, urinary net acid excretion, urinary bicarbonate and urinary ammonia.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients
* Age 21-75 years
* Six months since the time of the most recent transplant
* Serum bicarbonate 20-28mM on the two most recent serum measures with the last six months
* Stable creatinine

Exclusion Criteria:

* Systolic blood pressure > 140mmHg
* Diastolic blood pressure > 90mmHg
* Known ejection fraction <50%
* Clinical diagnosis of heart failure
* Use of >3 antihypertensive agents
* > 1+ edema
* Use of alkali in the preceding 3 months
* History of noncompliance with clinic visits

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Urinary transforming growth factor-beta1 | 6 months
  This is considered a surrogate marker of chronic allograft nephropathy (tubulointerstitial fibrosis).

SECONDARY OUTCOMES:
urinary ammonia excretion | 6 months
  a component of urinary acid excretion

CONTACTS AND LOCATIONS:
Overall Officials: Kalani L Raphael, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] de Brito-Ashurst I, Varagunam M, Raftery MJ, Yaqoob MM. Bicarbonate supplementation slows progression of CKD and improves nutritional status. J Am Soc Nephrol. 2009 Sep;20(9):2075-84. doi: 10.1681/ASN.2008111205. Epub 2009 Jul 16. PMID 19608703
- [Background] Amara AB, Sharma A, Alexander JL, Alfirevic A, Mohiuddin A, Pirmohamed M, Close GL, Grime S, Maltby P, Shawki H, Heyworth S, Shenkin A, Smith L, Sharma AK, Hammad A, Rustom R. Randomized controlled trial: lisinopril reduces proteinuria, ammonia, and renal polypeptide tubular catabolism in patients with chronic allograft nephropathy. Transplantation. 2010 Jan 15;89(1):104-14. doi: 10.1097/TP.0b013e3181bf13d9. PMID 20061926
- [Background] Mahajan A, Simoni J, Sheather SJ, Broglio KR, Rajab MH, Wesson DE. Daily oral sodium bicarbonate preserves glomerular filtration rate by slowing its decline in early hypertensive nephropathy. Kidney Int. 2010 Aug;78(3):303-9. doi: 10.1038/ki.2010.129. Epub 2010 May 5. PMID 20445497
- [Background] Raphael KL, Wei G, Baird BC, Greene T, Beddhu S. Higher serum bicarbonate levels within the normal range are associated with better survival and renal outcomes in African Americans. Kidney Int. 2011 Feb;79(3):356-62. doi: 10.1038/ki.2010.388. Epub 2010 Oct 20. PMID 20962743